CLINICAL TRIAL: NCT03939208
Title: Efficacy of a Brief Intervention Strategy for School Mental Health Clinicians (BRISC)
Brief Title: Efficacy of a Brief Intervention for School Clinicians (BRISC)
Acronym: BRISC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: Institute of Education Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Eric Bruns, Professor, School of Medicine: Psychiatry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 52229; R305A160111 (Other Grant/Funding Number: Institute of Education Sciences)
Record Dates: First submitted 2019-04-24; First posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Emotional/Behavioral Function; Academic Performance
Keywords: children's mental health; school mental health; evidence-based practice (EBP); academic success

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants include students, parents, and clinicians. Students and parents are prevented from having knowledge of the interventions assigned. Clinicians are aware of their intervention assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (BRISC) Group (Experimental): Clinicians randomly assigned to BRISC will implement a flexible intervention that, over four sessions, aims to assess and engage student clients, and identify and address student identified difficulties that are distressing and impacting academic performance/behavior, social, and overall functioning. BRISC uses an explicit, problem-solving structure and a range of techniques common to evidence-based practices (EBP) tailored to the identified needs of the student.
  Interventions: Behavioral: BRISC
- Services as Usual (SAU) Group (Active Comparator): Clinicians in the SAU condition will use a diverse array of "treatment as usual" strategies over four sessions that may include some directive, skill-building techniques common in EBPs, but, given findings from pilot studies and studies of mental health services "as usual" in community and school settings, are likely to be provided at an overall lower rate, and at lower intensity, than in BRISC or other EBP.
  Interventions: Behavioral: SAU

INTERVENTIONS:
Behavioral: BRISC
  Arms: Intervention (BRISC) Group
Behavioral: SAU
  Arms: Services as Usual (SAU) Group

SUMMARY:
Research shows that the majority of all mental health (MH) treatment for children is delivered in schools. Unfortunately, however, school mental health (SMH) providers rarely use evidence-based approaches and are often poorly integrated into the school context. Given the high (>20%) and increasing rates of MH disorders among children and youth, MH clinicians working in schools need effective and efficient ways to address student emotional and behavioral problems. The Brief Intervention Strategy for School Clinicians (BRISC) is a four-session, flexible, and research-informed "Tier 2" intervention tailored to high school students and designed to fit the school context. Findings from initial research funded by an IES Development and Innovation grant, including a small (n=66) comparison study, indicate positive, small to large sized effects (ES = .30- 1.33) in favor of BRISC for MH impairment, emotional symptoms, therapeutic alliance, coping skills, and client satisfaction. Moreover, even though the majority of students who were referred to BRISC were in the clinical range for functional impairment due to MH problems, over 50% were able to step down to lower levels of intervention after four sessions of BRISC, demonstrating promise for efficiency and reach. Given potential for public health impact, the purpose of the current study is to further examine the efficacy of BRISC by assessing its impact on mental health and academic outcomes - as well as feasibility, acceptability, and efficiency - in a larger, multi-site trial.

DETAILED DESCRIPTION:
Fostering emotional and behavioral well-being is critical to school success, and research shows that over 70% of all mental health treatment for children is delivered in schools. Thus, school mental health (SMH) services are a fundamental component of our nation's strategy to ensure academic and life success of our children and youth. Unfortunately, SMH providers rarely use evidence-based approaches and are often poorly integrated into the school context. SMH providers carry large caseloads, experience time constraints, and serve youth with a broad array of needs. For SMH to live up to its potential, individuals who provide SMH treatment must be equipped with effective and efficient ways to address student emotional and behavioral needs.

The purpose of this project is to conduct a multi-site randomized controlled trial (RCT) of the Brief Intervention Strategy for School Clinicians (BRISC). BRISC is a fully developed, manualized intervention strategy for use by professionals working individually with high school students experiencing mental health symptoms or other emotional and behavioral stressors that negatively affect their ability to succeed academically. With funding from an IES Development and Innovation grant (R305A120128), BRISC was developed as a brief, evidence-based, and flexible "Tier 2" intervention designed to fit the high school context. Findings from a small (N=66) comparison study indicate positive, small to large sized effects (ES = .30 - 1.33) in favor of BRISC over SMH services as usual (SAU) for a range of short and longer-term outcomes (see Section A9). The study also found high clinician fidelity to BRISC, increased clinician use of evidence-based strategies, high ratings of feasibility, and very low ratings of research burden. Moreover, even though the majority of students who were referred to BRISC were in the clinical range for functional impairment due to MH problems, over 50% were able to step down to lower levels of intervention after four sessions of BRISC, demonstrating promise for efficiency and reach. The current study aims to further examine the efficacy of BRISC, the mediators and moderators that may further influence its development, and to illuminate how and under what conditions BRISC is effective. A cluster randomized design has been used to assign 52 schools in Washington, Minnesota, and Maryland to BRISC or SAU (520 students total; 260 per group).

This efficacy project has six research aims:

1. To test the effects of BRISC on hypothesized short-term service outcomes such as clinician use of evidence-based strategies and standardized assessment data, therapeutic alliance, student service satisfaction, retention in services, and service referrals.
2. To test the effects of BRISC on hypothesized short-term student outcomes, such as problem-solving, coping skills, school engagement, school attendance, and homework completion.
3. To test the effects of BRISC on longer-term outcomes such as MH symptoms, emotional/behavioral functioning, peer/family relations, discipline problems at school, and academic performance.
4. To examine the impact of BRISC on treatment efficiency, in terms of trajectory of student change in outcomes over time.
5. To confirm that BRISC is perceived as an appropriate, feasible, and acceptable intervention for use by SMH clinicians working in a diverse array of high schools.
6. To examine hypothesized moderators and mediators of outcomes, including service factors (e.g., fidelity, service dosage/duration, clinician orientation, receipt of other services), student factors (e.g., age, gender, problem type and severity), and proximal outcomes (e.g., problem-solving skills, coping strategies, school engagement).

ELIGIBILITY:
Clinicians

Inclusion Criteria:

* SMH clinicians from a MH provider agency dedicated at .50 FTE to MH treatment (to ensure adequate integration in the school and students for the study) OR school counselors who are employed by the school district
* SMH clinicians or school counselors not currently receiving support to implement another specific intervention model
* Master's or Ph.D.-level mental health counselors

Exclusion Criteria:

- SMH clinicians with previous BRISC exposure

Students

Inclusion Criteria:

* Students must be age 14-21 years and enrolled in high school
* Students who are seeking or referred to services for the first time in the current school year, to minimize confusion about for which service episode measures should be completed
* English must be the first or primary language of the students
* If student is under 18 years old, a parent or legal guardian must consent for the student to participate

Exclusion Criteria:

* Students receiving Special Education services due to cognitive disability, due to inappropriateness of BRISC for youth with these disorders
* Students in foster care, due to challenges in obtaining consent to participate from public child welfare systems who serve as guardians
* Students who present currently in a crisis situation (defer to clinician's clinical judgment)

Parents/Guardians

Inclusion Criteria:

* Biological parent or legal guardian
* Must be English or Spanish speaking.

Exclusion Criteria:

- Parents who only speak any languages other than English or Spanish

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Internal and External Symptoms | Pre-intervention/baseline, 2-week follow-up, post-intervention/2 months, 4-month follow-up, 6-month follow-up
  The Brief Problem Checklist (BPC) is a youth/parent 12-item questionnaire adapted from items on the CBCL (Child Behavior Checklist) and YSR (Youth Self Report) designed to assess internalizing and externalizing behaviors with items measured on 0-2 scale. Subscale and total scores are mean scores of items with a range of 0-2. Higher scores reflect less favorable outcomes.
Change in Symptoms of Depression | Pre-intervention/baseline, post-intervention/2 months, 6-month follow-up
  The Patient Health Questionnaire (PHQ-9) is a widely-used, brief 9-item scale that queries about the presence depressive disorder symptoms with items on a 0-3 scale. Total scores are summed scores of items with a range of 0-27. Higher scores reflect more severe levels of depression.
Change in Symptoms of Anxiety | Pre-intervention/baseline, post-intervention/2 months, 6-month follow-up
  The Generalized Anxiety Disorder scale (GAD-7) is a widely-used, brief 7-item scale that queries about anxiety symptoms with items on a 0-3 scale. Total scores are summed scores of items with a range of 0-21. Higher scores reflect more severe levels of anxiety.
Change in Overall Mental Health Function | Pre-intervention/baseline, post-intervention/2 months, 6-month follow-up
  The Columbia Impairment Scale (CIS) is a 13-item scale that measures adolescents' level of adaptive functioning with items on a 0-4 scale. Total scores are summed scores of items with a range of 0-52. Higher scores reflect less favorable outcomes.

SECONDARY OUTCOMES:
Change in School Engagement | Pre-intervention/baseline, post-intervention/2 months, 6-month follow-up
  The Student Engagement Instrument (SEI) is a widely-used 35-item instrument that assesses engagement, a malleable determinant of high school success, with items on a scale of 0-3. SEI yields scores on six factors: teacher-student relationships, control and relevance of school work, peer support for learning, future aspirations and goals, family, support for learning, and extrinsic reward. Subscale and total scores are averaged scores of items with a range of 0-3. Higher scores reflect better outcomes.
Youth Satisfaction with Services | 2-month follow-up after baseline
  The Multidimensional Adolescent Satisfaction Scale (MASS) is a 21-item measure of client satisfaction with the services they receive from their mental health provider. The MASS includes four factors: counselor qualities, meeting needs, effectiveness, and counselor conflict. Items are on a 1-4 scale. Subscale and total scores are averaged scores of items with a range of 0-4. Higher scores reflect higher satisfaction with services.
Therapeutic Alliance | 2-month follow-up after baseline
  The Therapeutic Alliance Scale for Adolescents (TASA) is a widely used, 12-item scale designed to measure the working alliance between clinicians and their adolescent clients with items on a 1-6 scale. The scale covers three domains: bond, goals, and tasks. Subscale and total scores are averaged scores of items with a range of 1-6. Higher scores reflect better alliance.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington School Mental Health Assessment, Research, and Training (SMART) Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No